CLINICAL TRIAL: NCT01554735
Title: The Effects of Lifestyle-modification Induced Weight Loss on Metabolic and Inflammatory Profile, Endothelial, Sexual and Urinary Function, and Quality of Life in Obese Men
Brief Title: Effects of Lifestyle-modification Induced Weight Loss on Sexual and Urinary Function, and Quality of Life in Obese Men
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12200233
Record Dates: First submitted 2012-03-01; First posted 2012-03-15 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Sexual Dysfunction; Endothelial Dysfunction; Quality of Life; Inflammation
Keywords: obesity; men; sexual function; urinary tract symptoms; endothelial function; inflammation; quality of life
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Inflammation; Obesity; Multiple Endocrine Neoplasia Type 1 | interventions — Exercise; Diet; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lifestyle counselling (Experimental): exercise and diet counselling for weight loss
  Interventions: Behavioral: Exercise and diet

INTERVENTIONS:
Behavioral: Exercise and diet — 24 weeks of exercise and diet counselling
  Other Names: Diet advice; Exercise training

SUMMARY:
This study aims to evaluate the extent to which weight loss of 5-10% from baseline, induced by exercise and diet, improves metabolic and inflammatory profile, endothelial function, erectile function, sexual desire, lower urinary tract symptoms (LUTS), and quality of life in obese men.

DETAILED DESCRIPTION:
This study aims to evaluate the extent to which weight loss of 5-10% from baseline, induced by exercise and diet, improves metabolic and inflammatory profile, endothelial function, erectile function, sexual desire, lower urinary tract symptoms (LUTS), and quality of life in obese men.Men aged 30-65 years, with body mass index (BMI) ≥ 27.5 kg/m2, will be recruited from referrals to the Sports Medicine Centre in Changi General Hospital. The study will be conducted at the Sports Medicine Centre by trained medical investigators, dieticians and sports trainers.At baseline, 12 and 24 weeks, fasting glucose and lipids, insulin, testosterone, sex-hormone binding globulin, serum C-reactive protein and interleukin-6 are measured, endothelial function is measured by the non-invasive EndoPAT method, and validated questionnaires administered to assess changes in erectile function, sexual desire, LUTS and quality of life

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 30-65 years
* Body Mass Index (BMI) >/= 27.5 kg/m2
* Waist circumference (WC) >/= 90 cm

Exclusion Criteria:

* pituitary disease or cranial radiotherapy
* previous or current androgen replacement or deprivation therapy
* current treatment for sexual problems or LUTS
* glomerular filtration rate < 60 ml/min
* liver disease
* alcohol intake exceeding 500 g/week in the previous 12 months
* use of opiates, glucocorticoids, recreational drugs or phosphodiesterase inhibitors

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
erectile function | 24 weeks
  Increase in IIEF-5 score

SECONDARY OUTCOMES:
lower urinary tract symptoms | 24 weeks
  decrease in IPSS score

CONTACTS AND LOCATIONS:
Overall Officials: Joan J Khoo, MRCP, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Khoo J, Tian HH, Tan B, Chew K, Ng CS, Leong D, Teo RC, Chen RY. Comparing effects of low- and high-volume moderate-intensity exercise on sexual function and testosterone in obese men. J Sex Med. 2013 Jul;10(7):1823-32. doi: 10.1111/jsm.12154. Epub 2013 May 1. PMID 23635309